CLINICAL TRIAL: NCT03623347
Title: Neo-adjuvant Treatment of Glioblastomas With Marked to Severe Neurological Impairment Using Upfront Bevacizumab/témozolomide Association Before an Eventual Radiotherapy. Multicentric Phase II Study
Brief Title: Upfront Bevacizumab/témozolomide for Gliomastomas With Neurological Impairment
Acronym: TEMOBEVA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2011_843_0001
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2018-08

CONDITIONS: Chemoradiotherapy
Keywords: bully glioblastoma; multifocal glioblastoma; bevacizumab; temozolomide
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: TMZ and BEV induction before chemoradiotherapy — New approaches are needed for patients newly diagnosed with bulky glioblastoma (GB) and/or with severe neurological impairment that cannot benefit from first line temozolomide (TMZ)-based chemoradiotherapy.

SUMMARY:
New approaches are needed for patients newly diagnosed with bulky glioblastoma (GB) and/or with severe neurological impairment that cannot benefit from first line temozolomide (TMZ)-basedn chemoradiotherapy. Bevacizumab (BEV), an antiangiogenic anti-VEGF-R monoclonal antibody, has a rapid impact on tumor-related brain edema in recurrent GB. The present study reports the feasibility and efficacy of an induction treatment with TMZ and BEV to alleviate the initial neurological impairment and/or to reduce the tumor volume before a delayed chemoradiotherapy.

DETAILED DESCRIPTION:
New approaches are needed for patients newly diagnosed with bulky glioblastoma (GB) and/or with severe neurological impairment that cannot benefit from first line temozolomide (TMZ)-based chemoradiotherapy. Bevacizumab (BEV), an antiangiogenic anti-VEGF-R monoclonal antibody, has a rapid impact on tumor-related brain edema in recurrent GB. The present study reports the feasibility and efficacy of an induction treatment with TMZ and BEV to alleviate the initial neurological impairment and/or to reduce the tumor volume before a delayed chemoradiotherapy.

The investigators retrospectively analyzed tumor and target volumes and clinical neurological status in 39 patients with bulky GB and/or with severe neurological impairment after an induction treatment combining TMZ and BEV. Neurological and radiological responses were assessed according to RANO criteria.

Calculating gross tumor and clinical target volumes (GTV and CTV) was done at diagnosis and before radiotherapy. Progression-free survival (PFS) and overall survival (OS) were determined by Kaplan Meier methods. Safety was reported according to NCTCAE.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria:- - age> to 18 years

  * GBM de novo
  * Histological evidence is essential. A minimum interval of 7 days is required between biopsy and neo-adjuvant therapy. A minimum interval of 15 days is required for open skull surgery and neo-adjuvant therapy.
  * The insertion of patients is a WHO score 3 and 4 in relation to the neurological deficit is possible by definition
* Biological criteria

  - Polynuclear neutrophils> 1500 / mm3
  * pads> 100,000 / mm3
  * SGOT <5 at the upper limit of normal (ULN)
  * bilirubin <1.5 x ULN
  * Creatinine <1.5 ULN
  * proteinuria <2 g / 24 hours
* Forensic criteria

  * Patient with health insurance
  * consent signed by the patient if it is lucid, or by default by the person of trust.

Exclusion Criteria:

* 1. Patients without neurological deficit (SN 0) or with moderate deficit (SN 1 or SN 2).

  2. In case of initial neurological deficit SN 3-4, the interest of a decompression surgery must be discussed. If the surgery is unsuccessful, a corticosteroid test, at least 4 days, with at least 1.5 mg / kg / day of prednisone equivalent, must be performed. If surgery and / or corticosteroids allow to return to an SN 0-2 neurological score with return to an RPA III, IV or V class, the patient is not included and must be treated according to a conventional chemoradiotherapy regimen with temozolomide (Stupp schema).

  3. Multifocal tumor or whose excessive volume does not allow to consider curative radiation therapy at a dose of 60 Gy.

  3. History of chemotherapy, (including Gliadel) and / or radiotherapy. 4. Cerebral or intratumoral haemorrhage on diagnostic MRI. However, microhemorrhages, haemosiderin deposits or haemorrhages secondary to biopsy or surgery are not contraindications.

  5. Concomitant serious uncontrolled pathology, including another evolving cancer 6. Uncontrolled infection 7. Uncontrolled Hypertension (PAS> 160 mm Hg) Despite Optimized Treatment 8. Coronary artery disease or unstable arterial disease. Evolutionary aneurysm. Myocardial infarction less than 6 months old.

  9. Stroke or peripheral arterial disease less than 6 months old. 10. Heart Failure> NYHA Grade II 11. Haemorrhagiparous disease (hemophilia, Willebrandt ...) 12. History of hemoptysis less than 1 month old. 13. Pulmonary embolism less than 1 month old. 14. Anticoagulant or antiplatelet therapy in progress. If possible, these treatments should be stopped before inclusion after consultation with a cardiologist or angiologist. However, these treatments may be continued if their discontinuation is considered harmful and that the participation in the trial is considered beneficial for the patient with regard to the haemorrhagic risk incurred.

  15. Surgical procedure (other than craniotomy or stereotactic biopsy) less than one month old or foreseeable surgery.

  16. History of digestive fistula or intestinal perforation whose resolution is less than 6 months old.

  17. Pregnant or lactating patient (contraception to be prescribed if necessary) 18. Known intolerance to bevacizumab or temozolomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators retrospectively collected clinical and radiological data from medical files. Patients were over 18 years old. Most had histologically proven unresectable primary GB. in some cases, GB diagnosis was only done by multimodal MRI with confirmation by a collegial agreement including an expert in neuroradiology.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Optimal chemoradiotherapy after upfront TMZ and BEV treatment. | 4-months
  The investigators reported here a series of patients in whom radiotherapy was considered as not feasible in first intention but most of which could be treated by optimal chemoradiotherapy after upfront TMZ and BEV treatment. The investigators analyzed the impact of this induction strategy on tumor and target volumes, neurological status and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Boone, MD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No